CLINICAL TRIAL: NCT00881413
Title: Clinical Effectiveness of Intravenous Esomeprazole Versus Pantoprazole in Preventing Peptic Ulcer Recurrent Bleeding: a Double-Blind Randomized Trial
Brief Title: Esomeprazole Versus Pantoprazole to Prevent Peptic Ulcer Rebleeding
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: problems in funding
Sponsor: Lotung Poh-Ai Hospital (Other)
Collaborators: Tomorrow Medical Foundation (Other)
Responsible Party: Professor Hwai-Jeng Lin, Lotung Poh-Ai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMCP98004
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Peptic Ulcer
Keywords: Peptic ulcer bleeding; Proton pump inhibitor; Esomeprazole; Pantoprazole; Recurrent bleeding; bleeding
MeSH Terms: conditions — Peptic Ulcer; Peptic Ulcer Hemorrhage; Hemorrhage | interventions — Esomeprazole; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esomeprazole (Experimental): High-dose esomeprazole
  Interventions: Drug: Esomeprazole
- Pantoprazole (Active Comparator): High-dose pantoprazole
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Esomeprazole — Intravenous esomeprazole (Nexium®, AstraZeneca, Sodertalje, Sweden) is administered with 80mg bolus and 8mg/hr infusion for 72 hours. After 3 days, patients receive oral esomeprazole 40 mg (Nexium®, AstraZeneca, Sodertalje, Sweden) for 2 months
  Other Names: Nexium
  Arms: Esomeprazole
Drug: Pantoprazole — After successful endoscopy, intravenous pantoprazole (Pantoloc®, Nycomed GMBH, Konstanz, Germany) is administered with 80mg bolus and 8mg/hr infusion for 72 hours. After 3 days, patients receive oral pantoprazole 40 mg (Pantoloc®, Nycomed GMBH, Oranienburg, Germany) for 2 months
  Other Names: Pantoloc
  Arms: Pantoprazole

SUMMARY:
The aim of this study is to compare the clinical effectiveness of intravenous esomeprazole and pantoprazole in preventing recurrent bleeding in the patients with high-risk bleeding peptic ulcers after successful standard endoscopic hemostasis.

DETAILED DESCRIPTION:
Endoscopic hemostasis and proton pump inhibitor (PPI) constitute the cornerstone in the management of peptic ulcer bleeding (PUB), which remains a prevalent disorder associated with substantial morbidity and mortality. Clinical effectiveness of PPI in the management of patients with PUB has been established by compelling evidence derived from a number of randomized trials. However, whether different PPIs are equally effective has not been investigated. Esomeprazole, the S-isomer of omeprazole, may achieve faster, more profound and steady acid suppression than other PPIs, but it remains undetermined whether the superiority of pharmacologic efficacy may be translated into advantages in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years
* undergo emergent endoscopy within 24 hours of presentation
* have peptic ulcers in the gastroesophageal junction, stomach, or duodenum
* high-risk stigmata of peptic ulcers: Forrest classification IA~IIB
* endoscopic hemostasis by thermocoagulation or clip placement

Exclusion Criteria:

* pregnant or lactating
* written informed consent not obtained
* initial endoscopic hemostasis fail
* bleeding tendency (platelet count < 50×109/L, prolonged prothrombin time for more than 3 seconds, or were taking anticoagulants)
* PPI use within 14 days of enrollment
* comorbid with severe hepatic or renal insufficiency (serum total bilirubin more than 5 mg/dL, serum creatinine more than 5 mg/dL, or under dialysis)
* bleeding gastric cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
recurrent bleeding within 14 days of enrollment | 14 days after enrollment

SECONDARY OUTCOMES:
Volume of blood transfusion | 14 days after enrollment
Need for surgery | 14 days after enrollment
all-cause mortality | 14 days after enrollment
bleeding-related mortality | 14 days after enrollment
length of hospital stay | probably one month after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Hwai-Jeng Lin, M.D., Principal Investigator — Lotung Poh-Ai Hospital

REFERENCES:
- [Background] Sung JJ, Barkun A, Kuipers EJ, Mossner J, Jensen DM, Stuart R, Lau JY, Ahlbom H, Kilhamn J, Lind T; Peptic Ulcer Bleed Study Group. Intravenous esomeprazole for prevention of recurrent peptic ulcer bleeding: a randomized trial. Ann Intern Med. 2009 Apr 7;150(7):455-64. doi: 10.7326/0003-4819-150-7-200904070-00105. Epub 2009 Feb 16. PMID 19221370